CLINICAL TRIAL: NCT06582589
Title: Efficacy and Safety of Healsea® Children Isotonic Nasal Spray in the Prevention of Upper Respiratory Tract Infections With Nasal Symptoms in Children: a Pre-market Study
Brief Title: HEALSea Nasal Spray for Prevention of Infections in Children
Acronym: HEALSPIC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lallemand Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LPH-2402; 2819/02.08.2024 (Other: Republic of Bulgaria-Ministry of Health- Ethics Committe for Clinical Trials)
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Healthy Subjects
Keywords: Prevention; Nasal spray; upper respiratory tract infection; saline solution
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Prospective randomized open label pre-market clinical investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healsea Children treated group (Experimental): Subjects of this arm will be treated with Healsea Children nasal spray (1 puff in each nostril twice daily) during 3 treatment periods of 28 days interspersed by 2 wash-out periods of 10 days
  Interventions: Device: Healsea Children
- untreated group (No Intervention): Subjects of this arm will not receive any treatment for the prevention of respiratory tract infection.

INTERVENTIONS:
Device: Healsea Children — Subjects will use Healsea Children 1 puff in each nostril twice daily upon awakening and at bedtime, during three 28-day treatment periods interspersed by a 10-day wash-out
  Arms: Healsea Children treated group

SUMMARY:
Healsea® Children is a class IIa medical device. This is an isotonic seawater-based nasal spray supplemented with a natural Symbiofilm™ extract (0.02%) isolated from marine bacteria. Healsea® Children is indicated in children above 6 years to clean and moisten the nose during colds.

Symbiofilm™, which is not a medicinal product is able to protect the nasal mucosa from viruses' entrance by forming a protective barrier on the nasal mucosa.

By targeting the nose as entry points for viruses, we hypothesise that Healsea® Children used regularly during the respiratory virus season may prevent upper respiratory tracts infections such as cold or flu with nasal symptoms.

The main objective of this premarket clinical investigation is thus to assess the efficacy of Healsea® Children to prevent upper respiratory tract infections with nasal symptoms in healthy children during 3 treatment periods of 28 days interspersed by 2 wash-out periods of 10 days when compared to children not taking Healsea® Children.

138 children will be randomised in the study, 64 in the Healsea® Children group and 64 in the non-treated group.

The subjects (or their parents) will be asked to report the upper respiratory tract infections with nasal symptoms and complication they may have during the study to the physician in charge of the study conduct.

Two study visits and 3 telephone calls are scheduled. The subjects will also complete an electronic diary to report nasal symptoms and adverse event other than upper respiratory tracts infections.

DETAILED DESCRIPTION:
Upper respiratory tract infections (URTIs) and sino-nasal symptoms are very frequent.

Human rhinovirus (more than 100 serotypes) is the most common cause, accounting up to 50% viral rhinitis episodes in children and adults. These episodes can last up to 7-10 days and are usually self-limited. Prevalence of acute rhinosinusitis varies with season (higher in the fall and winter months) and climatic variations and increases with a damp environment and air pollution. It is estimated that an infant can typically have up to 11 upper respiratory tract infection episodes per year with URTIs being one of the main causes of primary care consultations. The number usually diminishes with age, with generally around eight episodes at preschool age and four at school age.

Healsea® Children is a class IIa medical device. This is an isotonic seawater-based nasal spray supplemented with a natural Symbiofilm™ extract (0.02%) isolated from marine bacteria. Healsea® Children is indicated in children above 6 years to clean and moisten the nose during colds and rhinitis. The clinical performance of Healsea® Children is supported by the sea water solution and Symbiofilm™. The exact mechanisms by which nasal irrigation works are not known. However, most of the experts agree that it is primarily a mechanical intervention leading to direct cleaning of the nasal mucosa.

The other component of Healsea® Children, Symbiofilm™ is an exopolymeric composition with emulsifying/surfactant properties which enhance the cleansing and moistening of nasal mucosa. Furthermore, a prophylactic activity of Symbiofilm™ against infection by viruses involved in upper respiratory infections i.e., Adenovirus, Rhinovirus, Flu virus and OC 43 Coronavirus has been demonstrated in vitro on human nasal epithelial cells (HNEpC). The antiviral prophylactic activity of Symbiofilm™ is suggested to rely on its physiochemical properties that, by coating the surface of epithelial cells, hinders the viral entry process, thus explaining the reduced viral adsorption and the subsequent reduced onset of infection.

By targeting the nose as entry points for viruses, we hypothesise that Healsea® Children used regularly during the respiratory virus season may prevent upper respiratory tracts infections with nasal symptoms.

The aim of this two arms prospective randomized open-labelled pre-market clinical investigation, is to establish clinical benefits and clinical safety of Healsea® Children to prevent upper respiratory tract infections with nasal symptoms in healthy children during 3 treatment periods of 28 days (one puff in each ostril twice daily) interspersed by 2 wash-out periods of 10 days when compared to children not taking Healsea® Children.

138 children will be randomised in the study, 64 in the Healsea® Children group and 64 in the non-treated group.

The subjects (or their parents) will be asked to immediately call the investigator in case of nasal symptoms and complication of respiratory infection they may have during the study.

Two study visits (Visit 1, Screening/Randomisation at Day 1 and Visit 2, End of study visit at Day 106 up to Day 116) and 3 telephone calls (telephone call 1 TC1 at Day15 ±3 days, TC2 at Day 55 ±3 days and TC3 at Day 95±3days) are scheduled. The subjects will also complete an electronic diary to report nasal symptoms, device deficiencies, and adverse events other than upper respiratory tracts infections from D2 up to end of study (Day 106 up to Day 116).

The duration of patient's participation is up to 116 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female subjects ≥6 and <18-year-old
2. No respiratory tract infection within 15 days before trial entry and at trial entry
3. Written consent obtained from parent/legal guardians
4. Written assent obtained from patient
5. Availability of a smartphone throughout the study and an internet connection.-

Exclusion Criteria:

1. Known hypersensitivity/allergy to any component of the test device,
2. Subject with severe asthma, perennial allergy, cystic fibrosis, immunodeficiency or ciliary dyskinesis,
3. Body temperature ≥ 37.5°
4. Medical history or any current disease that is considered by the investigator as a reason for non-inclusion,
5. Severe nasal septum deviation or other condition that could cause nasal obstruction such as the presence of nasal polyps,
6. Antibiotic (systemic or per nasal route) or antivirals (systemic) intake within 2 weeks before screening,
7. Systemic or local corticosteroids (nasal route or inhalation) within 4 weeks before screening,
8. Antihistamines intake for allergy when treatment was started from less than 4 weeks before screening,
9. Vaccination against flu or COVID-19 within 6 months before screening,
10. Chronic decongestant use within 2 weeks before screening,
11. Bacterial lysates or immunostimulants (food supplements excluded) used for prevention of infection within the 6 months before the screening,
12. Prebiotics, probiotics used for prevention of infection within 6 months before the screening,
13. Pregnant/Lactating female or with sexual activity without hormonal contraception, intrauterine device or barrier methods.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 139 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects without any upper respiratory tract infection (URTI) with nasal symptoms during the study. | From the randomization up to Day 116
  The upper respiratory tracts infections with nasal symptoms (blocked nose, runny nose yellow or green discharge, sneezing ) will be collected for each subject throughout An URTI episode with nasal symptoms is defined as follows: (i) at least 1 of the followings must be present: a blocked nose, runny nose, yellow or green nasal discharge, sneezing; (ii) the symptomatic episode must last for at least 3 days.

SECONDARY OUTCOMES:
Time to first Upper Respiratory Tract Infection with nasal symptoms during the study | From the randomization up to Day 116
  The time to first Upper Respiratory Tract Infection with nasal symptoms (blocked nose, runny nose, yellow or green discharge, sneezing) will be compared between groups
Number of Upper Respiratory Tract Infections with nasal symptoms during the study | From the randomization up to Day 116
  Upper Respiratory Tract Infections with nasal symptoms will be reported by the subjects to the investigators during the whole study duration and the total number compared between groups
Number of Upper Respiratory Tract Infections complications | From the randomization up to Day 116
  Complications of Upper respiratory Tract Infections (bronchitis, bronchiolitis, pneumoniae, pharyngo-tonsillitis, laryngitis, acute otitis) will be reported by the subjects during the whole study duration and compared between groups
Number of days of use of concomitant treatments that may affect Upper Respiratory Tract Infections symptoms and associated complications | From the randomization up to Day 116
  The number of days of antipyretics intake, systemic or local mucolytics, decongestants, antitussives, systemic and per nasal route antibiotics, local and systemic corticosteroids, systemic antivirals) will be compared between the 2 arms
Number of school days lost due to Upper Respiratory Tract Infections and complications | From the randomization up to Day 116
  Number of school days lost due to Upper Respiratory Tract Infections and complications will be collected during the whole study duration and compared between groups
Assessment of (serious) adverse events and device deficiences throughout the study | From the randomization up to Day 116

CONTACTS AND LOCATIONS:
Locations (8):
- Bulgaria (8):
  - Multiprofile Hospital for Active Treatment Sveti Ivan Rilski -2003 OOD, Dupnitsa
  - Medical Center Plovdimed Ltd, Plovdiv
  - Medical Center Iskar EOOD, Sofia
  - Medical Center Polymed AD, Sofia
  - Medical Center First Pediatric, Sofia
  - Multiprofile Hospital for active treatment, Sofia
  - Diagnostics and Consultation Center Convex EOOD, Sofia
  - Ambulatory for individual Practice for specialized outpatient medical care for children's diseases and pediatric pneumology ans phtysiatry, Vratsa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tano L, Tano K. A daily nasal spray with saline prevents symptoms of rhinitis. Acta Otolaryngol. 2004 Nov;124(9):1059-62. doi: 10.1080/00016480410017657. PMID 15513550
- [Background] Cabaillot A, Vorilhon P, Roca M, Boussageon R, Eschalier B, Pereirad B. Saline nasal irrigation for acute upper respiratory tract infections in infants and children: A systematic review and meta-analysis. Paediatr Respir Rev. 2020 Nov;36:151-158. doi: 10.1016/j.prrv.2019.11.003. Epub 2020 Feb 21. PMID 32312677
- [Background] Stanfel D, Kalogjera L, Ryazantsev SV, Hlaca K, Radtsig EY, Teimuraz R, Hrabac P. The Role of Seawater and Saline Solutions in Treatment of Upper Respiratory Conditions. Mar Drugs. 2022 May 17;20(5):330. doi: 10.3390/md20050330. PMID 35621981
- [Background] Slapak I, Skoupa J, Strnad P, Hornik P. Efficacy of isotonic nasal wash (seawater) in the treatment and prevention of rhinitis in children. Arch Otolaryngol Head Neck Surg. 2008 Jan;134(1):67-74. doi: 10.1001/archoto.2007.19. PMID 18209140
- [Background] Williamson S, Dennison L, Greenwell K, Denison-Day J, Mowbray F, Richards-Hall S, Smith D, Bradbury K, Ainsworth B, Little P, Geraghty AWA, Yardley L. Using nasal sprays to prevent respiratory tract infections: a qualitative study of online consumer reviews and primary care patient interviews. BMJ Open. 2022 Jun 30;12(6):e059661. doi: 10.1136/bmjopen-2021-059661. PMID 35772824